CLINICAL TRIAL: NCT05748587
Title: Role of Iron, Alpha-Synuclein, and Lymphocyte-activation Gene-3 in the Pathophysiology of Ischemic Stroke in Human and Albino Rats
Brief Title: Iron, Alpha-Synuclein, and Lymphocyte-activation Gene-3 in Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Asmaa Abdel-mageed Muhammed, Lecturer, Aswan University Hospital
Other Study IDs: sLAG-3 in brain ischemia
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Brain Ischemia
MeSH Terms: conditions — Brain Ischemia | interventions — Deferoxamine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control: 24 healthy age and sex-matched controls
  Interventions: Diagnostic Test: Serum Iron; Diagnostic Test: RBCs Alpha-synuclein; Diagnostic Test: Serum Soluble lymphocyte activation gene; Radiation: Brain computed tomography
- Patients with acute Ischemic stroke: 24 patients between 50-70 years having neurological symptoms of acute ischemic stroke will be included.
  Patients with acute hemorrhagic stroke, Parkinson's disease, dementia, Alzheimer's disease, malignancy, and central nervous system infection will be excluded.
  Interventions: Diagnostic Test: Serum Iron; Diagnostic Test: RBCs Alpha-synuclein; Diagnostic Test: Serum Soluble lymphocyte activation gene; Radiation: Brain computed tomography
- Control rats: 8 rats will be subjected to a Sham operation and will be injected intramuscularly immediately after the operation with an equivalent 0.9% saline solution. After 24 hours they will be sacrificed.
  Interventions: Diagnostic Test: Brain Iron; Diagnostic Test: Brain Alpha-synuclein; Diagnostic Test: Brain lymphocyte activation gene
- Rats with ischemic stroke: 8 rats will be subjected to bilateral common carotid artery occlusion (CCAO) for 30 minutes and will be injected intramuscularly immediately after removing the occlusion with an equivalent 0.9% saline solution. They will be sacrificed after 24 hours of reperfusion.
  Interventions: Diagnostic Test: Brain Iron; Diagnostic Test: Brain Alpha-synuclein; Diagnostic Test: Brain lymphocyte activation gene
- Rats with ischemic stroke + deferoxamine: 8 rats will be subjected to bilateral CCAO for 30 minutes and will be injected intramuscularly immediately after removing the occlusion with deferoxamine (200 mg/kg), They will be sacrificed after 24 hours of reperfusion.
  Interventions: Diagnostic Test: Brain Iron; Diagnostic Test: Brain Alpha-synuclein; Diagnostic Test: Brain lymphocyte activation gene; Drug: Deferoxamine

INTERVENTIONS:
Diagnostic Test: Serum Iron — Serum iron levels in study groups
  Groups: Control; Patients with acute Ischemic stroke
Diagnostic Test: RBCs Alpha-synuclein — α-syn levels in RBCs
  Other Names: α-syn
  Groups: Control; Patients with acute Ischemic stroke
Diagnostic Test: Serum Soluble lymphocyte activation gene — sLAG-3 in the serum of study groups
  Other Names: sLAG-3
  Groups: Control; Patients with acute Ischemic stroke
Radiation: Brain computed tomography — Brain CT of patients after admission
  Other Names: CT
  Groups: Control; Patients with acute Ischemic stroke
Diagnostic Test: Brain Iron — Iron in brain homogenate of rats
  Groups: Control rats; Rats with ischemic stroke; Rats with ischemic stroke + deferoxamine
Diagnostic Test: Brain Alpha-synuclein — α-syn expression in rat's brain
  Other Names: α-syn
  Groups: Control rats; Rats with ischemic stroke; Rats with ischemic stroke + deferoxamine
Diagnostic Test: Brain lymphocyte activation gene — LAG-3 expression in rat's brain
  Other Names: LAG-3
  Groups: Control rats; Rats with ischemic stroke; Rats with ischemic stroke + deferoxamine
Drug: Deferoxamine — intramuscular deferoxamine (200 mg/kg) injection to rats
  Groups: Rats with ischemic stroke + deferoxamine

SUMMARY:
This observational study aims to detect levels of iron, alpha-synuclein, and soluble lymphocyte activation gene 3 in acute ischemic stroke patients. And to see expressions of iron, alpha-synuclein, and lymphocyte activation gene 3 in the brain tissue of ischemic rats. The main questions it aims to answer are:

* Is there an association between iron and alpha-synuclein accumulation in ischemic stroke?
* Is there any change in soluble lymphocyte activation gene levels in ischemic stroke and if these levels are related to stroke severity and infarction size? . Can soluble lymphocyte activation gene levels be used as an early biomarker to diagnose ischemic stroke?

ELIGIBILITY:
Inclusion Criteria:

1. Patients at the age between 50-70 years.
2. Patients having neurological symptoms of acute ischemic stroke.

Exclusion Criteria:

1. Patients with acute hemorrhagic stroke.
2. Patients with Parkinson's disease (PD).
3. Patients with dementia, and Alzheimer's disease.
4. Patients with any type of malignancy.
5. Patients with central nervous system infection.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurological symptoms of acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Iron levels | 6 months
  Serum iron levels in ischemic patients and control
Alpha-synuclein levels | 6 months
  Alpha-synuclein levels in RBCs in ischemic patients and control
Levels of Soluble lymphocyte activation gene-3 | 6 months
  Serum soluble lymphocyte activation gene-3 in ischemic patients and control
levels of iron, alpha-synuclein, and soluble lymphocyte activation in relation to stroke severity and infarction size | 6 months
  stroke severity will be evaluated by the National Institutes of Health Stroke Scale (NIHSS) and size of infarction will be detected by brain CT
Iron levels in brain of rats | 2 months
  Iron levels in brain homogenate of rats in the three rat groups
Levels of Alpha-synuclein expression in brain of rats | 2 months
  Alpha-synuclein expression in brain of rats in different groups
Levels of Lymphocyte activation gene-3 expression in brain of rats | 2 months
  lymphocyte activation gene-3 expression in brain of rats in different groups

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Abdelmageed Muhammed, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt

REFERENCES:
- [Background] Malfertheiner K, Stefanova N, Heras-Garvin A. The Concept of alpha-Synuclein Strains and How Different Conformations May Explain Distinct Neurodegenerative Disorders. Front Neurol. 2021 Oct 5;12:737195. doi: 10.3389/fneur.2021.737195. eCollection 2021. PMID 34675870
- [Background] Wu Q, Wei C, Guo S, Liu J, Xiao H, Wu S, Wu B, Liu M. Acute iron overload aggravates blood-brain barrier disruption and hemorrhagic transformation after transient focal ischemia in rats with hyperglycemia. IBRO Neurosci Rep. 2022 Jul 3;13:87-95. doi: 10.1016/j.ibneur.2022.06.006. eCollection 2022 Dec. PMID 35847179
- [Background] Yoon CW, Park HK, Bae EK, Rha JH. Sleep Apnea and Early Neurological Deterioration in Acute Ischemic Stroke. J Stroke Cerebrovasc Dis. 2020 Feb;29(2):104510. doi: 10.1016/j.jstrokecerebrovasdis.2019.104510. Epub 2019 Nov 22. PMID 31767524
- [Background] Zhao L, Wang H, Xu K, Liu X, He Y. Update on lymphocyte-activation gene 3 (LAG-3) in cancers: from biological properties to clinical applications. Chin Med J (Engl). 2022 May 20;135(10):1203-1212. doi: 10.1097/CM9.0000000000001981. PMID 35170503